CLINICAL TRIAL: NCT02267512
Title: Efficacy and Safety of Two Anti-T-lymphocyte Immune Globulin (ATG-F) Induction Regimens in de Novo Kidney Transplant Patients - a Multicenter, Randomized, Parallel Group Study
Brief Title: Efficacy and Safety of Two Anti-T-lymphocyte Immune Globulin (ATG-F) Induction Regimens in Anew Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACN-ATG-KTx-12-1
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: De Novo Kidney Transplant Patients
Keywords: Kidney Transplant Patients; ATG-F

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATG-F single dosing group (Experimental): Intravenous (IV)
  Interventions: Drug: ATG-F
- ATG-F continuous dosing group (Experimental): Intravenous (IV)
  Interventions: Drug: ATG-F

INTERVENTIONS:
Drug: ATG-F — Intravenous (IV)

SUMMARY:
To investigate the efficacy and safety of ATG-F induction regimen using a single dose of ATG-F compared with a five-day dose regimen of ATG-F in anew kidney transplant recipients.

DETAILED DESCRIPTION:
To investigate the efficacy and safety of ATG-F induction regimen using a single dose of ATG-F compared with a five-day dose regimen of ATG-F in de novo kidney transplant recipients. The primary analysis of this study is to demonstrate the non-inferiority of the two regimens with regard to efficacy, defined as failure rate.

The secondary objective of the study is the assessment of safety and further efficacy parameters in terms of incidence of acute rejections, graft/patient survival, DGF(delayed graft function) and renal function

ELIGIBILITY:
Inclusion Criteria:

* Patient with end stage kidney disease who is a suitable candidate for primary kidney transplantation.
* Patients scheduled to undergo renal allograft transplantation with compatible ABO blood type.
* Peak PRA <50%
* Females of childbearing potential must have a negative pregnancy test within 48hrs prior to randomization and reliable methods of contraception should be started 4 weeks prior to and during the whole study.
* Patients capable to understand the purposes and risks of the study, who are willing and able to participate in the study and from whom written and dated informed consent to participate in the study is obtained.

Exclusion Criteria:

* Subject has previously received or is receiving an organ transplant other than kidney
* Subject is receiving double-kidney transplant.
* Subject is receiving an ABO incompatible or T-cells cross match positive transplant.
* Cold ischemia time of allograft is > 24 hours before kidney transplantation surgery.
* Subject is receiving organ from a Human Leukocyte Antibody (HLA) identical donor.
* Known contraindication to administration of ATG-F, including:

  * Subject has known hypersensitivity to rabbit proteins
  * Subject with severe thrombocytopenia
  * Subject with bacterial, viral or mycotic infections which are not under therapeutically control
* Subject has known hypersensitivity to tacrolimus, macrolide antibiotics, mycophenolate mofetil, or any of the product excipients.
* Subject is unlikely to comply with the visits scheduled in the protocol in the opinion of the investigator or has a history of non-compliance.
* Pregnant women, nursing mothers, lactating women, and women of child-bearing potential who are unwilling to use reliable contraception during the study and for 6 weeks following completion of the study.
* Patients with evidence of active liver disease (liver function tests ≥ 2 times upper limit of normal) or the presence of a chronic active hepatitis B or C.
* Recipient or donor is seropositive for human immunodeficiency virus (HIV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
efficacy failure | 12 months post-transplant
  Efficacy failure is defined as any of the following events:
  * patient's death,
  * graft loss,
  * acute rejection,
  * and/or lost to follow-up.

SECONDARY OUTCOMES:
Incidence of acute rejection | 6 and 12 months
Incidence of DGF | 6 and 12 months
  DGF = delayed graft function
Incidence of patient survival | 6 and 12 months
Incidence of graft survival | 6 and 12 months
Renal function: serum creatinine/eGFR | 1, 3, 6 and 12 months
incidence and severity of AEs | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (14):
- China (14):
  - Beijing
  - Changchun
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Jinan
  - Nanjing
  - Shanghai
  - Shenyang
  - Tianjin
  - Wenzhou
  - Wuhan
  - Xi'an
  - Zhengzhou

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=201